CLINICAL TRIAL: NCT00443872
Title: Adding Orally Disintegrating Selegiline (Zelapar) to Patients Taking Dopamine Agonists and Experiencing Complications
Brief Title: Efficacy of Orally Disintegrating Selegiline in Parkinson's Patients Experiencing Adverse Effects With Dopamine Agonists
Acronym: AtoZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parkinson's Disease and Movement Disorder Center of Boca Raton (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Stuart Isaacson, MD, Director of the Parkinson's Disease and Movement Disorder Center of Boca Raton, Parkinson's Disease and Movement Disorder Center of Boca Raton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAL-1.0-IV
Record Dates: First submitted 2007-03-03; First posted 2007-03-06 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Dopamine agonist adverse effects; MAO-B inhibitor; orally disintegrating selegiline; Zelapar
MeSH Terms: conditions — Parkinson Disease | interventions — Selegiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- orally disintegrating selegiline (Other): This is a one arm open label study of patients who are experiencing a dopamine agonist (DA) related adverse effects (AE) of either one or more of the following: excessive daytime sleepiness, hallucinations, pedal edema, impulse control disorder. All subjects received orally disintegrating selegiline.
  Interventions: Drug: orally disintegrating selegiline (Zelapar)

INTERVENTIONS:
Drug: orally disintegrating selegiline (Zelapar) — 1.25 mg once daily orally disintegrating selegiline for 6 weeks with an increase to 2.5 mg once daily orally disintegrating selegiline for remaining 6 weeks if tolerated

SUMMARY:
The purpose of the study is to determine if reducing or eliminating a dopamine agonist (DA) causing one of the side effects of daytime sleepiness, swelling of the lower legs or feet, hallucinations or impulsive behaviors while adding orally disintegrating selegiline can eliminate the adverse effect and maintain control of Parkinson's disease (PD) symptoms.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disease. Symptomatic therapy is primarily aimed at restoring dopamine function in the brain. Levodopa is the most effective symptomatic treatment; however, long term use is associated with motor fluctuations (periods of return of PD symptoms when medication effect wears off) and dyskinesia (drug induced involuntary movements including chorea and dystonia). Once patients develop motor fluctuations treatment options include increasing the frequency of levodopa dosing, switching to sustained-release levodopa, adding other therapies including monoamine oxidase type B (MAO-B) inhibitors, dopamine agonists, catechol-o-methyltransferase (COMT) inhibitors and in patients with severe motor fluctuations deep brain stimulation surgery. There are no good evidence based studies indicating whether the use of one of these class of drugs is superior to the other nor are there treatment algorithms that recommend which class of drug should be initiated when the patients initially develop motor fluctuations. It is believed that the efficacy of the different drug classes is similar. However, the frequency of adverse effects may differ between drug classes, but such studies are lacking. In clinical practice when patients develop adverse effects to a drug from one class, a drug from another class is substituted in an attempt to maintain efficacy with reduced adverse effects.

Dopamine agonists often have a higher risk of adverse effects compared to MAO B inhibitors. Therefore, the rationale for this study is that the addition of orally disintegrating selegiline after the reduction or discontinuation of the offending dopamine agonist will result in comparable efficacy with reduced adverse events. This study will assess the safety and efficacy of the addition of orally disintegrating selegiline in PD patients who are having adverse effects to dopamine agonists for which a dose reduction of the dopamine agonist is being considered. All patients in the study will receive orally disintegrating selegiline 1.25 mg once a day and the dose will be increased to 2.5 mg once a day if tolerated.

Comparisons: The status of the adverse event at the end of the study while on orally disintegrating selegiline will be compared to the adverse event at the start of the study. In addition, efficacy will be compared at the start of the study while on the dopamine agonist to the end of the study with orally disintegrating selegiline.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (PD) confirmed by at least two of the following signs: resting tremor, bradykinesia,rigidity
* Male or female outpatients
* Age 30-90 years
* Current use of levodopa (stable for at least 1 month) and a dopamine agonist (pramipexole or ropinirole)
* Treatment response to current anti-parkinsonian medications in the opinion of the investigator
* Dopamine agonist adverse effect that in the opinion of the investigator requires a reduction or discontinuation of the dopamine agonist. The adverse effects must be in one of the following four categories and should not be so severe as to require immediate discontinuation of the dopamine agonist (i.e., hallucinations without insight, serious impulsive behavior resulting in significant loss or danger to the patient).

Daytime sleepiness - must score >10 on Epworth Sleepiness Scale (ESS) at Baseline; Pedal edema - bothersome/concerning to patient; Hallucinations - insight should be maintained; Impulsive behavior - not including behaviors that are harmful to the patient requiring immediate discontinuation of the agonist.

* Daily off time
* Acceptable contraception for females of child bearing potential
* Willing and able to comply with study procedures.
* Willing and able to give written informed consent prior to beginning any study procedures.

Exclusion Criteria:

* Atypical parkinsonism due to drugs, metabolic disorders, encephalitis, trauma, or other neurodegenerative diseases.
* Significant cognitive or psychiatric impairment which, in the opinion of the investigator, would interfere with the ability to complete all the tests required in the protocol.
* Participation in another clinical drug trial within the previous four weeks.
* Patients currently on monoamine oxidase type A or B (MAO-A or B) inhibitors, meperidine, tramadol, methadone, propoxyphene, dextromethorphan, and mirtazapine.
* History of hypersensitivity or adverse reaction to selegiline or previous exposure to orally disintegrating selegiline
* History of melanoma
* Unstable/uncontrolled medical problems
* History of drug/alcohol abuse

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Pahwa, MD, Principal Investigator — University of Kansas Medical Center
Locations (17):
- United States (17):
  - University of California - Irvine, Irvine, California
  - Coastal Neurological Medical Group, Inc, La Jolla, California
  - University of Southern California, Los Angeles, California
  - The Parkinson's Institute, Sunnyvale, California
  - Parkinson's Disease and Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - University of South Florida, Tampa, Florida
  - Methodist Plaza Speciality Clinic, Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Henry Ford Health Center - Franklin Pointe, Southfield, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - University of Toledo, Toledo, Ohio
  - NeuroHealth Parkinson Disease and Movement Disorder Center, Warwick, Rhode Island
  - Neurology Specialists Dallas, Dallas, Texas
  - ETMC Neurological Institute, Tyler, Texas

REFERENCES:
- [Result] Lyons KE, Friedman JH, Hermanowicz N, Isaacson SH, Hauser RA, Hersh BP, Silver DE, Tetrud JW, Elmer LW, Parashos SA, Struck LK, Lew MF, Pahwa R. Orally disintegrating selegiline in Parkinson patients with dopamine agonist-related adverse effects. Clin Neuropharmacol. 2010 Jan-Feb;33(1):5-10. doi: 10.1097/WNF.0b013e3181b7926f. PMID 19855267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parkinson's disease (PD) patients with levodopa-induced motor fluctuations were enrolled at 12 sites in the United States. The first subject was enrolled in March 2007, and the last subject completed in September 2008.
Pre-assignment Details: Excessive daytime sleepiness was defined by an Epworth Sleepiness Scale (ESS) score greater than 10; pedal edema was bothersome to the subject; hallucinations were bothersome, but insight was maintained; and impulse control disorders (ICDs) included behaviors not requiring immediate medical attention and not harmful to the patient or to others.
Groups:
- PD Patients With DA Related AE: This is a one arm open label study of PD patients with a DA related AE
Period: Overall Study
Arm/Group | PD Patients With DA Related AE
Started | 77
Completed | 60
Not Completed | 17
Not completed — Protocol Violation | 7
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 8

BASELINE CHARACTERISTICS:
Arm/Group | PD Patients With DA Related AE
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Reduction in Adverse Events
Description: The primary outcome measure was the reduction of daytime sleepiness, hallucinations, pedal edema, and impulse control disorders after a reduction of dopamine agonist dose with the addition of an monoamine oxidase (MAO)-B inhibitor (orally disintegrating selegiline). Percentages of participants with reduction in individual adverse events as well as reduction in any adverse events are reported.
Time Frame: 3 Months
Population: 77 patients enrolled in the study and 60 completed. Each patient had to have at least one of the following DA related AEs, excessive daytime sleepiness, hallucinations, pedal edema or impulse control disorder (they could have more than one AE). 60 subjects were selected based on results of previous studies (discontinued patients were replaced).
Measure: Number; unit: percentage of participants
Groups:
- PD Patients With DA Related AE: Patients who are experiencing a dopamine agonist (DA) related adverse effect (AE) of either one or more of the following: excessive daytime sleepiness, hallucinations, pedal edema, impulse control disorder, received 1.25 mg once daily orally disintegrating selegiline for 6 weeks with an increase to 2.5 mg once daily orally disintegrating selegiline for remaining 6 weeks if tolerated.
Arm/Group | PD Patients With DA Related AE
Number analyzed (Participants) | 60
percentage of participants
  Excessive Daytime Sleepiness (n=50) | 94
  Hallucinations (n=15) | 86
  Pedal Edema (n=26) | 73
  Impulse Control Disorder (n=25) | 84
  Any Adverse Event (n=60) | 100

2. Primary Outcome: Epworth Sleepiness Scale Score for Those With Daytime Sleepiness
Description: This is a measure of daytime sleepiness. The test is a list of eight situations in which one rates their tendency to become sleepy on a scale of 0, no change of dozing to 3, high chance of dozing. The total score ranges fro 0-24, with higher values representing excessive sleepiness. A score of greater than 10 represents clinically significant sleepiness.
Time Frame: Baseline and 3 months
Population: Based only on the number of patients with excessive daytime sleepiness at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PD Patients With DA Related AE (Daytime Sleepiness): Patients who are experiencing a dopamine agonist (DA) related adverse effect (AE) of daytime sleepiness received 1.25 mg once daily of orally disintegrating selegiline for 6 weeks with an increase to 2.5 mg once daily orally disintegrating selegiline for the remaining 6 weeks if tolerated.
Arm/Group | PD Patients With DA Related AE (Daytime Sleepiness)
Number analyzed (Participants) | 50
units on a scale
  Baseline | 13.5 (3.0)
  3 months (12 weeks) | 9.0 (3.7)
Statistical Analysis 1: Comparison: PD Patients With DA Related AE (Daytime Sleepiness); Comparison of mean group scores at baseline and 12 weeks; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 4.5, Standard Deviation 1

3. Primary Outcome: Neuropsychiatric Inventory (NPI) Hallucinations Scale Score for Those With Hallucinations
Description: Report of hallucinations with insight maintained based on the hallucinations questions of the Neuropsychiatric Inventory (NPI). The participant and their caregiver are asked a series of questions to determine if hallucinations are present. If present they rate the frequency of hallucinations on a scale of 1 (rarely, less than once a week) to 4, very often (once or more daily). They also rate the severity of the hallucinations, as mild (1 - present but harmless and cause little distress), moderate (2 - distressing and disruptive) or severe (3 - very disruptive, major source of behavioral disturbance, may need meds). The frequency and severity scores are multiplied (maximum score 12, with higher scores representing more distress/disability) for the total score.
Time Frame: Baseline and 3 months
Population: Patients who reported hallucinations at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PD Patients With DA Related AE (Hallucinations): Patients who are experiencing the dopamine agonist (DA) related adverse effect of hallucinations. The participants received 1.25 mg once daily of orally disintegrating selegiline for 6 weeks after which it was increased to 2.5 mg once daily if tolerated.
Arm/Group | PD Patients With DA Related AE (Hallucinations)
Number analyzed (Participants) | 15
units on a scale
  Baseline | 3.3 (2.7)
  3 months (12 weeks) | 1.3 (1.8)
Statistical Analysis 1: Comparison: PD Patients With DA Related AE (Hallucinations); Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.0

4. Primary Outcome: Circumference of Lower Leg/Foot at Greatest Point of Swelling for Pedal Edema
Description: The circumference of the lower leg/ankle with the greatest swelling was measured using a standard tape measure at baseline and 12 weeks for both the right and left ankles.
Time Frame: Baseline and 3 months
Population: Presence of pedal edema at baseline
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- PD Patiens With DA Related AE (Pedal Edema): Patients who are experiencing a dopamine agonist (DA) related AE of pedal edema received 1.25mg once daily of orally disintegrating selegiline for 6 weeks after which there was an increase to 2.5 mg once daily if tolerated.
Arm/Group | PD Patiens With DA Related AE (Pedal Edema)
Number analyzed (Participants) | 26
centimeters
  Left foot baseline | 25.8 (3.4)
  Left foot 3 months (12 weeks) | 24.6 (3.1)
  Right foot baseline | 26.4 (4.2)
  Right Foot 3 months (12 weeks) | 25.2 (4.0)
Statistical Analysis 1: Comparison: PD Patiens With DA Related AE (Pedal Edema); Change in pedal edema as measured by change in lower leg/ankle circumference in the left and right legs; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 1.2 — Comparison of baseline vs. 3 month circumference of the Left and Right lower leg/ankle (change identical for both legs)

5. Primary Outcome: Barratt Impulsiveness Scale Score for Those With Impulsive Behavior
Description: This is a measure of impulsiveness. There are 30 questions regarding the presence of impulsive and non-impulsive behaviors each scored from 1 (rarely/never) to 4 (almost always/always). The total score reflects the sum of the 30 items. A higher score represents more impulsiveness.
Time Frame: Baseline and 3 months
Population: The number with ICDs at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PD Patients With DA Related AE (Impulse Control Disorder): Patients who are experiencing dopamine agonist (DA) related adverse effect (AE) of impulse control disorder (ICD) received 1.25 mg once daily of orally disintegrating selegiline for 6 weeks after which it was increased to 2.5mg once daily if tolerated.
Arm/Group | PD Patients With DA Related AE (Impulse Control Disorder)
Number analyzed (Participants) | 25
units on a scale
  Baseline | 64.1 (11.4)
  3 months (12 weeks) | 61.3 (12.4)
Statistical Analysis 1: Comparison: PD Patients With DA Related AE (Impulse Control Disorder); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.8

6. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Scores
Description: The UPDRS activities of daily living sub scale has 14 questions regarding the ability to perform daily activities like dressing, eating, etc. These questions are completed by the patient and each question has 5 responses ranging from 0 (no problems) to 4 (severe disability/cannot do). The total score for this sub scale is the sum of the scores for the 14 questions (higher scores represent greater disability), maximum score is 56.
  The motor assessment is completed by the investigator. There are 14 questions evaluating motor function in various body parts, representing 27 individual items (i.e., some questions, such as rigidity, are rated for 5 different body parts, other questions, such as finger tapping, are rated on both the right and left sides, and other questions are rated individually). Each item has 5 responses, 0 being none/no disability and 4 being the most severe disability. The 27 items are summed (higher scores represent greater disability); maximum score is 108.
Time Frame: Baseline and 3 months
Population: All subjects completing the study were included
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Subjects With DA Related AEs (UPDRS Data): For all completed subjects (60) UPDRS activities of daily living scores and motor scores were collected. All patients received 1.25 mg once daily orally disintegrating selegiline for 6 weeks which was increased to 2.5mg once daily at 12 weeks if tolerated.
Arm/Group | All Subjects With DA Related AEs (UPDRS Data)
Number analyzed (Participants) | 60
units on a scale
  ADLs baseline | 11.9 (5.8)
  ADLs 3 months (12 weeks) | 10.3 (5.1)
  Motor baseline | 23.6 (10.9)
  Motor 3 months (12 weeks) | 21.4 (10.4)
Statistical Analysis 1: Comparison: All Subjects With DA Related AEs (UPDRS Data); This analysis is for the Activities of Daily Living (ADL) section of the scale; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.6
Statistical Analysis 2: Comparison: All Subjects With DA Related AEs (UPDRS Data); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — This analysis is for the motor section of the UPDRS; Mean Difference (Final Values) = 2.2

7. Secondary Outcome: PDQ-39 Quality of Life Assessment Total Scores
Description: The PDQ-39 is a measure of quality of life, it has 8 sub scales and a total score. For this study only the total score was examined. There are a total of 39 questions related to the following 8 sub scales: ability/difficulty to perform motor activities, ability to perform daily activities, cognition, emotional well being, stigma, social support, communication, bodily discomfort; each question with 5 responses (0, no/never, 4 always). The total score is calculated by adding the scores for each of the 39 items, dividing by 39 x 4 (maximum score for all 39 items) and then multiplying by 100 to get a percentage score ranging from 0-100 with 100 representing the most disability and greatest impact on quality of life.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Subjects PDQ-39: This includes all patients in the study. They all received 1.25 mg once daily of orally disintegrating selegiline for 6 weeks which was increased to 2.5 mg once daily if tolerated.
Arm/Group | All Subjects PDQ-39
Number analyzed (Participants) | 60
units on a scale
  Baseline | 28.6 (15.3)
  3 months (12 weeks) | 24.4 (15.1)
Statistical Analysis 1: Comparison: All Subjects PDQ-39; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 4.2

8. Secondary Outcome: Beck Depression Inventory for All Subjects
Description: The Beck Depression Inventory is a general measure of depression. There are 21 questions each with responses ranging from 0 (no issue or problem) to 3 (maximum issue/distress), all questions are related to emotions, mood, feelings, etc. The total possible score is 63 (higher scores represent more depression). The total score is calculated by adding the scores of the 21 items.
Time Frame: Baseline and 3 months
Population: All
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All PD Patients With DA Related AEs (BDI): All patients had a DA related AE and received 1.25 mg once daily orally disintegrating selegiline which was increased after 6 weeks to 2.5mg once daily if tolerated.
Arm/Group | All PD Patients With DA Related AEs (BDI)
Number analyzed (Participants) | 60
units on a scale
  Baseline | 10.2 (6.4)
  3 months (12 weeks) | 9.4 (7.4)
Statistical Analysis 1: Comparison: All PD Patients With DA Related AEs (BDI); Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.8

9. Secondary Outcome: Beck Anxiety Inventory Scores for All Subjects
Description: The Beck Anxiety Inventory is a general measure of anxiety. There are 21 questions each with responses ranging from 0 (no issue or problem) to 3 (severe - I could barely stand it), all questions are related to the presence of signs or symptoms of anxiety. The total possible score is 63 and a higher score represents greater anxiety. The total score is calculated by adding the responses for each of the 21 items.
Time Frame: Baseline and 3 months
Population: All
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All PD Patients With DA Related AEs (BAI): All patients had a DA related AE and received 1.25 mg once daily orally disintegrating selegiline which was increased after 6 weeks to 2.5mg once daily if tolerated.
Arm/Group | All PD Patients With DA Related AEs (BAI)
Number analyzed (Participants) | 60
units on a scale
  Baseline | 11.5 (9.7)
  3 months (12 weeks) | 10.9 (10.2)
Statistical Analysis 1: Comparison: All PD Patients With DA Related AEs (BAI); Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.6

10. Secondary Outcome: Mini Mental State Examination (MMSE) Scores for All Subjects
Description: The MMSE is a general measure of cognition (i.e., measures attention, memory, visuospatial construction, etc). It has 30 items, each item representing 1 point. The total score ranges from 0-30 with 30 being a perfect score (no cognitive impairment) and 0 being the lowest score (greatest possible level of impairment). The total score is calculated by adding the scores of each item.
Time Frame: Baseline and 3 months
Population: All
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All PD Patients With DA Related AEs (MMSE): All patients had a DA related AE and received 1.25 mg once daily orally disintegrating selegiline which was increased after 6 weeks to 2.5mg once daily if tolerated.
Arm/Group | All PD Patients With DA Related AEs (MMSE)
Number analyzed (Participants) | 60
units on a scale
  Baseline | 28.8 (1.6)
  3 months (12 weeks) | 29.2 (1.2)
Statistical Analysis 1: Comparison: All PD Patients With DA Related AEs (MMSE); Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.4

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | PD Patients With DA Related AE
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 57/77
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD Patients With DA Related AE (N=77)
worsening of PD (Nervous system disorders) | 13 (13)
Nausea/vomiting (Gastrointestinal disorders) | 11 (11)
Dyskinesia (Nervous system disorders) | 8 (8)
Increased body aches and pain (General disorders) | 6 (6)
Increased insomnia (General disorders) | 5 (5)
Increased anxiety (Psychiatric disorders) | 4 (4)
Restless legs (Nervous system disorders) | 4 (4)
orthostatic hypotension (Cardiac disorders) | 4 (4)
Increased depression (Psychiatric disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No